CLINICAL TRIAL: NCT03561532
Title: FECAL MICROBIOTA TRANSPLANTATION IN THE TREATMENT OF ULCERATIVE COLITIS
Brief Title: Fecal Transplantation in Ulcerative Colitis
Acronym: FMT-CU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Helsinki University Central Hospital (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUS / 1652/2016
Record Dates: First submitted 2018-06-06; First posted 2018-06-19 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Participants are randomized in two groups to receive in colonoscopy either a fecal suspension made of their own feces or a fecal suspension of a healthy donor.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant and the treating personnel are blinded of the randomization result.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT (Active Comparator): 50% of the participants will receive fecal suspension of a healthy donor administered in colonoscopy into the cecum
  Interventions: Other: Fecal microbiota transplantation (FMT)
- Placebo (Placebo Comparator): 50% of the participants will receive fecal suspension made of their own feces administered in colonoscopy into the cecum.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fecal microbiota transplantation (FMT) — FMT administered into the cecum of the patient in colonoscopy.
  Arms: FMT
Other: Placebo — Autologous FMT (fecal suspension made of patients own feces) administered into the cecum of the patient in colonoscopy.
  Arms: Placebo

SUMMARY:
Adult individuals with ulcerative colitis in remission are given a single fecal microbiota transplantation (FMT) in colonoscopy. A half of the patients will receive autologous FMT as a placebo and a half will receive an FMT from a healthy donor.

DETAILED DESCRIPTION:
80 adult patients with ulcerative colitis (UC) will be recruited. They are randomized to receive either an autologous FMT as a placebo or FMT from a healthy donor (frozen and thawed).

The patients are followed up with fecal samples to detect microbial changes. The follow up lasts 1 year after the FMT and a follow up colonoscopy will be done 52 weeks after the FMT.

ELIGIBILITY:
Inclusion Criteria:

* • • Diagnosis of CU based on clinical, endoscopic, and histological findings.

  * Remission assessed by Mayo score (0 to 1) and F-Calpro (<100 ug/g).
  * Availability of consecutive fecal samples during one year after the diagnosis of CU.
  * Availability of blood sample to study the IBD associated genetic background
  * Compliance to attend ileocolonoscopy and FMT within 3-6 months after the diagnosis of CU and at 52 week
  * 18-75 years

Exclusion Criteria:

* Unable to provide informed consent
* Need for any antibiotic therapy within 3 months
* Use of corticosteroids, immunosuppressive or biological medication at the baseline
* Use of any probiotics
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Maintenance of remission of ulcerative colitis | 52 weeks
  Endoscopic remission and Mayo-score < 2

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Päijät-Häme Central Hospital, Lahti

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.